CLINICAL TRIAL: NCT04380714
Title: Changes in the Consumption of Psychoactive Substances by People Incarcerated at the Villeneuve-Lès-Maguelone Prison During Containment Linked to COVID-19.
Brief Title: Changes in the Consumption of Psychoactive Substances During Containment Linked to COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0273
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: People Incarcerated; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SARS-CoV 2 pandemic started in China in December 2019, then reached France on January 24, 2020.

On March 14, France moved into phase 3 of the epidemic threshold with the implementation of containment measures on March 17 Measures were put in place by N.Belloubet (French Minister of Justice) from March 17, including suspension of visiting rooms and activities in detention.

Containment provides boredom and isolation with many potential consequences: sleep disturbance, anxiety, PTSD, depression, suicide, addictive behavior and violence.

However,prisoners have a higher prevalence of substance use disorders than the general population.

What will have been the impact of the confinement on the consumption of psychoactive substances by prisoners at the Villeneuve Les Maguelone prison.

* Anonymous questionnaire from the start
* Collection of socio-demographic data
* Collection of consumption data before and during containment
* Collection of monitoring data

ELIGIBILITY:
Inclusion criteria:

* Men incarcerated at Villeneuve Les Maguelone prison
* On a given date (May 12)
* Major
* French speaking
* non illiterate

Exclusion criteria:

* minors
* patients refusing
* non-French speaking
* illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People incarcerated in Villeneuve-Lès-Maguelon prison
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
percentage changes in the consumption of psychoactive substances | 1 day
  percentage changes in the consumption of psychoactive substances

SECONDARY OUTCOMES:
Assessment of the level of stress | 1 day
  Assessment of the level of stress by self-administered questionnaire before / during confinement
Assessment of depression | 1 day
  Assessment of depression by self-administered questionnaire before / during confinement
Craving modification evaluation | 1 day
  Craving modification evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Mieuset, PhD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC